CLINICAL TRIAL: NCT05368064
Title: Cleidocranial Dysplasia (CCD): From Genotype to Phenotype and Considerations for Care
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Greenberg Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00246592
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Cleidocranial Dysostosis
MeSH Terms: conditions — Cleidocranial Dysplasia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood or saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — collection of phenotype data

SUMMARY:
Cleidocranial Dysplasia (CCD) is a rare, autosomal dominant disorder characterized by dysplasia of bones and teeth. Given the rarity of this condition (prevalence of 1 in 1,000,000), the variable phenotype and lack of correlation to specific genotypes, coordinated clinical research is needed to better understand CCD. The purpose of this project is to: investigate the genetic makeup and phenotypic expression of CCD, understand the quality of life for patients with this diagnosis, and further identify the multidimensional healthcare needs of these patients. Participation involves completion of a survey to ascertain medical history and quality of life, a physical exam and research whole exome sequencing from a blood or saliva sample. The goal of this research is to elucidate critical pathways in skeletal and dental development and improve quality of life for CCD patients through the standardization and optimization of timely diagnosis and multidisciplinary care.

ELIGIBILITY:
Inclusion Criteria:

* Patient has molecular or clinical diagnosis of CCD
* Caregiver or parent of patient with CCD.

Exclusion Criteria:

* Patient does not have CCD
* Patient over 18 but cannot consent for themselves
* Not fluent in English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with clinical or molecular diagnosis of CCD
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of RUNX2 mutation | 3 years
  identify the RUNX2 mutation in each participant
Phenotypic description of each patient with CCD | 3 years
  Physical exam, dental exam, medical history collection

SECONDARY OUTCOMES:
Patient financial stress quality of life score as assessed by the Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT) | 3 years
  Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT) will be used to assess financial quality of life stress; numeric response 0-4; Score range 0-44 with higher scores indicating better Financial Well-Being.
Patient-reported health-related quality of life as assessed by the FANLTC (Functional Assessment of Non-life-threatening conditions) | 3 years
  FAN LTC (0 = not al all, 4 = very much)
Patient-reported health-related quality of life | 3 years
  Quality of Life questionnaire (7 = delighted, 1 = terrible)
Caregiver-reported quality of life of caregivers for patients with CCD | 3 years
  COST-FACIT (variable quality of numeric response 0-4); FAN LTC (0 = not at all, 4 = very much)
Whole exome sequencing if RUNX2 molecular analysis negative for pathogenic variant | 3 years
  sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Ickow, DMD, MS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided